CLINICAL TRIAL: NCT06265987
Title: ECHOQUALITY2: Maternal and Fetal Characteristics Influencing Image Quality in Prenatal Ultrasonography
Brief Title: Maternal and Fetal Characteristics Influencing Image Quality in Prenatal Ultrasonography
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECHOQUALITY2
Record Dates: First submitted 2024-02-03; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ultrasonography; Obstetrics; Fetus; Pregnant Women
Keywords: Quality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational study is to identify maternal and fetal characteristics that impact image quality in prenatal ultrasonography. The investigators have assembled a retrospective cohort of 198 patients, each contributing three ultrasound images taken between 18 and 18 weeks and 6 days of gestation. For each image, the investigators assess the quality of two distinct elements as well as the overall image through both subjective and objective evaluations.

The primary questions the study seeks to address are:

What maternal and fetal characteristics influence image quality in prenatal ultrasonography?

ELIGIBILITY:
Inclusion Criteria:

- Patient who underwent ultrasound between 18 weeks and 18 weeks + 6 days for prenatal diagnosis

* Ultrasound performed by the same practitioner
* Ultrasound performed on the same ultrasound machine "Voluson E10", with the "RM6C" probe

Exclusion Criteria:

- Patient's refusal

* Use of another ultrasound device other than the "Voluson E10", and/or an ultrasound probe other than the "RM6C"
* Intrauterine fetal deaths

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women having undergone an ultrasound between 18 weeks and 18 weeks + 6 days at the Multidisciplinary Prenatal Diagnostic Center of Poitiers University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Maternal and fetal characteristics can influence quality image in ultrasonography | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital La MILETRIE, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided